CLINICAL TRIAL: NCT06528145
Title: Comparison of Quality of Life and Functional Capacity of Long Covid Patients and Symptom-Free Volunteers: a Randomized Controlled Study
Brief Title: Long Covid (Individuals with Ongoing COVID-19 Symptoms) Ongoing Effects
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Ziya Yildiz (Other)
Collaborators: Suleyman Demirel University (Other); Pamukkale University (Other)
Responsible Party: Sponsor-Investigator, Ziya Yildiz, Dr. PhD (physiotherapy and rehabilitation), Isparta University of Applied Sciences
Organization: Isparta University of Applied Sciences (Other)
Other Study IDs: SülDemirelUni_YildizA_002
Record Dates: First submitted 2024-07-29; First posted 2024-07-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 Infection
Keywords: Long Covid; Quality of Life; COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- S-: Individuals who have not had symptoms for 6-18 months after Covid infection
  Interventions: Other: Evalation
- S+: Individuals with ongoing symptoms 6-18 months after Covid infection
  Interventions: Other: Evalation

INTERVENTIONS:
Other: Evalation — Post Covid Functional Scale (PCFS) was used to assess the functional status of the participants; Short Form- 36 (SF-36) questionnaire was used to assess quality of life; 30 s sit-to-stand test (30s-STS) and 6 min walk test (6 MWT) were used to assess functional capacity.

SUMMARY:
Persistent Covid-19 symptoms, known as long Covid, can impact healthcare provision. This study aimed to assess how symptoms persisting six months after Covid-19 affect quality of life and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* The study included individuals who had Covid-19 disease at least 6-18 months ago, who agreed to participate, and who were diagnosed with Covid-19 by a health institu-tion during the disease period.

Exclusion Criteria:

* Individuals who were not between the ages of 18-65, who had cognitive and commu-nicative impairments, and who had orthopedic and neurological limitations that would prevent them from performing physical activity were excluded from the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had an infection at Süleyman Demirel University Hospital at least 6 and up to 18 months ago and were re-admitted to the hospital due to symptoms were included.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Functional capacity, physical function, physical role difficulties, emotional role difficulties, pain and general health | 1 year
  Functional capacity was affected more in the group whose symptoms persisted than in the group whose symptoms did not persist (p<0.05). Some of the SF-36 sub-parameters (physical function, physical role difficulties, emotional role difficulties, pain and general health) were found to be sig-nificantly more affected in participants with persistent symptoms (p<0.05).

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Univesity, Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided